CLINICAL TRIAL: NCT01530984
Title: Anti-CTLA4 Blockade Alone or Combined With Systemic GM-CSF for Prostate Cancer Immunotherapy
Brief Title: Ipilimumab and GMCSF Immunotherapy for Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to execute contract
Sponsor: Lawrence Fong (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Lawrence Fong, Associate Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC# 12552
Record Dates: First submitted 2012-02-07; First posted 2012-02-10 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; metastatic castrate resistant prostate cancer; Chemotherapy-naïve patients; Anti-CTLA4 blockade; systemic GM-CSF; Ipilimumab
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ipilimumab alone (Experimental): Ipilimumab 3 mg/kg (IV) will be given every 28 days for six cycles (induction) followed by administration once every three months for patients who are not progressing (maintenance).
  Interventions: Drug: Ipilimumab
- Ipilimumab with GM-CSF (Experimental): Ipilimumab 3 mg/kg (IV) will be given every 28 days for six cycles (induction) followed by administration once every three months for patients who are not progressing (maintenance). GM-CSF 250 mcg/m2 SQ will be administered on days 1-14 in Cycles 1-6 and then every 3 months for 14 days beginning on the day of ipilimumab administration during the maintenance therapy phase
  Interventions: Drug: Ipilimumab; Drug: GM-CSF

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 3 mg/kg on day 1 of a 28 day cycle for 6 cycles.
  Other Names: CTLA-4 blockade
Drug: GM-CSF — GM-CSF 250 mcg/m2 SQ on days 1-14 for 6 cycles.
  Other Names: Sargramostim
  Arms: Ipilimumab with GM-CSF

SUMMARY:
This is an open-label randomized phase II study. Patients are randomized so as to achieve uniform patient cohorts treated on each regimen. Twenty-seven patients will be required per treatment arm, and a total of 54 prostate cancer patients will be required to complete this study. The study will assess for clinical activity by Prostate Specific Antigen (PSA) response, of both single agent ipilimumab and the combination of GM-CSF and ipilimumab in chemotherapy-naïve patients with metastatic castrate resistant prostate cancer.

DETAILED DESCRIPTION:
Ipilimumab is an antibody (proteins that can find and destroy foreign molecules such as those on bacteria and viruses) against CTLA-4 (a molecule that controls a part of the immune system by shutting it down). It is approved by the U.S. Food and Drug Administration (FDA) to treat patients with late-stage melanoma, skin cancer. The use of ipilimumab in patients with CRPC has not been approved by the FDA.

Some patients in this study will receive GM-CSF along with ipilimumab. In clinical trials, GM-CSF has been safely given to prostate cancer patients in combination with ipilimumab. GM-CSF is not approved by the FDA for use as treatment for prostate cancer. Studies in patients with prostate cancer suggest that GM-CSF may activate the immune system. Since ipilimumab can help keep the immune system from turning off and allow an immune reaction to occur, and GM-CSF can increase the activity of the immune system, it is possible that they may work together to increase the immune response to cancer. The use of ipilimumab in combination with GM-CSF in patients with CRPC has not been approved by the FDA.

It is theorized that if antigen presentation could be improved, the immunostimulatory effects of CTLA-4 blockade could be augmented with improvements in clinical response. To that end, UCSF conducted a phase I clinical trial of ipilimumab in combination with GM-CSF, a cytokine that has been demonstrated to enhance the functional activities of effector cells, including dendritic cells (DC), neutrophils, and monocytes, in chemotherapy-naïve men with CRPC (Protocol 6032).32 Exposure to GM-CSF increases class II MHC expression on dendritic cells and is thought to lead to increased antigen presentation to T cells, stimulating T cell responses, although this mechanism has not been confirmed. We have extensively studied the effects of treatment demonstrating a dose-response relationship in the activation of CD4 and CD8 T cells. Moreover, the expansion of activated (CD25+CD69+) CD4 and CD8 T cells seen with this GM-CSF/ipilimumab combination trial was higher than that seen with GM-CSF or ipilimumab monotherapy seen in our other trials in prostate cancer patients.

We are proposing to conduct a non-comparative randomized phase II study of repetitive dosing of ipilimumab either alone or in combination with GM-CSF in patients with metastatic CRPC. The dosing interval for ipilimumab is based on the prior study which demonstrated drug levels ≥ 10 mg/mL (a minimum level required for CTLA-4 blockade in pre-clinical models) for greater than 28 days. Six doses of ipilimumab were chosen because six doses have been given safely in other trials. Maintenance dosing every three months is empirical, but this dosing frequency is based on discussions with Medarex, Inc. and Bristol-Meyers Squibb and is based on reports indicating the safety and potential efficacy of this maintenance regimen.

This study will use ipilimumab given every 28 days for six cycles (induction) followed by administration once every three months for patients who are not progressing (maintenance). A dosage of 10 mg/kg has been chosen based on the results to date of the phase I study. GM-CSF 250 mcg/m2 SQ will be administered on days 1-14 in Cycles 1-6 and then every 3 months for 14 days beginning on the day of ipilimumab administration during the maintenance therapy phase.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, metastatic prostate cancer (positive bone scan and/or measurable disease on CT scan and/or MRI of the abdomen and pelvis).
2. Progressive disease after androgen deprivation, as defined by PSA Working Group 237 and/or RECIST criteria.38 Patients must have disease progression by one or both of the following:

   * For patients with measurable disease, progression is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions or the appearance of one or more new lesions, as per RECIST criteria version 1.1
   * For patients with no measurable disease, a positive bone scan and elevated PSA will be required. PSA evidence for progressive prostate cancer consists of a PSA level of at least 2 ng/ml, which has risen on at least 2 successive occasions, at least 1 week apart. If the confirmatory PSA (#3) value is not greater (i.e., #3b) than the screening PSA (#2) value, then an additional test for rising PSA (#4) will be required to document progression
   * If no prior orchiectomy has been performed, patients must remain on LHRH agonist or antagonist therapy. Patients who are receiving an antiandrogen as part of primary androgen ablation must demonstrate disease progression following discontinuation of the antiandrogen, defined as two consecutive rising PSA values, obtained at least two weeks apart, or documented osseous or soft tissue progression. At least one of the PSA values must be obtained at least four weeks (flutamide) or six weeks (bicalutamide or nilutamide) after discontinuation
3. Laboratory requirements:

   * Absolute neutrophil count (ANC) ≥ 1500/μL
   * Bilirubin < 1.5 x ULN
   * Hemoglobin ≥ 8 g/dL
   * PSA ≥ 2 ng/mL
   * Platelets > 100,000/μL
   * AST and ALT < 2.5 x ULN
   * Creatinine clearance ≥ 60mL/min by the Cockcroft Gault equation Testosterone < 50 ng/dL
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2 and life expectancy > 12 weeks.
5. At least 18 years of age or older.
6. Patients receiving any other hormonal therapy, including any dose of megestrol acetate (Megace), Proscar (finasteride), any herbal product known to decrease PSA levels (e.g. Saw Palmetto, PC-SPES), or any systemic corticosteroid, must discontinue the agent for at least four weeks prior to study treatment. Progressive disease as defined above must be documented after discontinuation of any hormonal therapy (with the exception of a LHRH agonist or antagonist).
7. Prior radiation therapy must be completed > 4 weeks prior to enrollment and the patient must be recovered from all toxicity. Prior radiopharmaceuticals (strontium, samarium) must be completed ≥ 8 weeks prior to enrollment.
8. Because of the unknown potential risk to a gamete and/or developing embryo from this investigational therapy, patients must agree to use adequate contraception (barrier method for males) for the duration of study participation, and for three months after discontinuing therapy.

Exclusion Criteria:

1. Prior chemotherapy for prostate cancer, with the exception of neoadjuvant chemotherapy, because of the potential effect of chemotherapy on the immune system.
2. Prior investigational immunotherapy. Prior sipuleucel-T treatment is allowed but must be completed at least 4 weeks prior to initiating treatment on this protocol.
3. Current treatment with systemic steroid therapy (inhaled/topical steroids are acceptable). Systemic corticosteroids must be discontinued for at least 4 weeks prior to first treatment.
4. History of autoimmune disease including, but not limited to:

   * Systemic lupus erythematosis (SLE), scleroderma, CREST syndrome, rheumatoid arthritis
   * Inflammatory bowel disease, celiac disease, primary biliary cirrhosis, autoimmune hepatitis
   * Dermatomyositis, polymyositis, giant cell arteritis
   * Autoimmune hemolytic anemia (AIHA), cryoglobulinemia, antiphospholipid antibody syndrome (APLS)
   * Diabetes mellitus type I, myasthenia gravis, Grave's disease
   * Wegener's granulomatosis or other vasculitis
   * A history of Hashimoto's thyroiditis, psoriasis, or eczema, any of which has been inactive for at least one year, or isolated Raynaud's phenomenon is acceptable
5. History or radiologic evidence of central nervous system metastases.
6. Medical or psychiatric illness that would preclude participation in the study or the ability of patients to provide informed consent for themselves.
7. Cardiovascular disease that meets one of the following: congestive heart failure (New York Heart Association Class III or IV), active angina pectoris, or recent myocardial infarction (within the last 6 months).
8. Concurrent or prior malignancy except for the following:

   * Adequately treated basal or squamous cell skin cancer
   * Adequately treated stage I or II cancer from which the patient is currently in complete remission
   * Any other cancer from which the patient has been disease-free for 5 years
9. HIV or other history of immunodeficiency disorder.
10. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or medical (e.g. infectious) illness.
11. Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
12. A history of prior treatment with ipilimumab or prior CD137 agonist or CTLA 4 inhibitor or agonist.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
To assess for clinical activity by PSA response, of both single agent ipilimumab and the combination of GM-CSF and ipilimumab in chemotherapy-naïve patients with metastatic castrate resistant prostate cancer. | 12 weeks
  To assess for clinical activity by PSA (prostate-specific antigen) decline of both single agent ipilimumab in chemotherapy-naïve patients with metastatic castrate resistant prostate cancer (CRPC). The primary endpoint is the proportion of treated patients achieving a >30% decline in PSA.

SECONDARY OUTCOMES:
To evaluate the duration of PSA response and time to PSA progression. To quantify the frequency of immune toxicities. To evaluate T cell activation. To assess for clinical activity by objective response. | 12 weeks

OTHER OUTCOMES:
Assessment of circulating tumor cell (CTC) frequency | 12 weeks
  To assess whether either treatment can modulate the frequency of circulating tumor cells (CTC). Modulation of the frequency of circulating tumor cells (CTC) will be measured from baseline to Cycle 6/off study visit of treatment.
Assessment of the antigen specific immune responses induced with treatment | 12 weeks
  Antigen specific immune responses will be measured by immunoblotting to detect the induction of IgG antibodies and by ELISA and ELISPOT assays to detect antibody and CD4 T cell responses, respectively, against candidate antigens in prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fong, MD, Principal Investigator — University of California, San Francisco; Lawrence Fong, MD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States